CLINICAL TRIAL: NCT02174718
Title: Evaluation of a Transdermal Vitamin D3 Delivery System, D3forME
Acronym: D3forME
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to manufacturing problems the transdermal patch was not produced.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0766
Record Dates: First submitted 2014-06-18; First posted 2014-06-25 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Vitamin D Deficiency
Keywords: Cholecalciferol; Transdermal patch
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Daily 4000IU transdermal D patch (Experimental): Only in the stage 2, Efficacy Study
  Interventions: Dietary Supplement: Transdermal D Patch
- Daily placebo patch plus oral placebo (Active Comparator): Only in the stage 3, non-inferiority Study
  Interventions: Dietary Supplement: Placebo patch; Dietary Supplement: Oral placebo
- Daily placebo patch plus oral vitamin D (Active Comparator): Only in the stage 3 Non-inferiority Study
  Interventions: Dietary Supplement: Oral vitamin D3; Dietary Supplement: Placebo patch
- Daily 4000IU topical patch plus oral placebo (Active Comparator): Only for the 3rd Stage of the study, Non-inferiority Study
  Interventions: Dietary Supplement: Transdermal D Patch; Dietary Supplement: Oral placebo
- Daily transdermal placebo patch (Placebo Comparator): Only in the stage 2, Efficacy Study
  Interventions: Dietary Supplement: Placebo patch

INTERVENTIONS:
Dietary Supplement: Transdermal D Patch
  Arms: Daily 4000IU topical patch plus oral placebo; Daily 4000IU transdermal D patch
Dietary Supplement: Oral vitamin D3
  Other Names: Obtained from Tischon corporation
  Arms: Daily placebo patch plus oral vitamin D
Dietary Supplement: Placebo patch
  Arms: Daily placebo patch plus oral placebo; Daily placebo patch plus oral vitamin D; Daily transdermal placebo patch
Dietary Supplement: Oral placebo
  Arms: Daily 4000IU topical patch plus oral placebo; Daily placebo patch plus oral placebo

SUMMARY:
A clinical need exists for non-oral vitamin D administration. This study is designed to test a new proprietary transdermal system. It is looking to see if this new system will safely and successfully deliver vitamin D3 to humans.

DETAILED DESCRIPTION:
This will be conducted in 3 stages. The hypotheses of this work are as follows:

1. The D3forME topical supplement patch will effectively and safely raise serum 25(OH)D3 in humans.
2. The 25(OH)D3 increment with a daily 4,000 IU D3forME topical supplement patch will be superior to a placebo patch.
3. The 25(OH)D3 increment with a daily 4,000 IU D3forME topical supplement patch will be non-inferior to that achieved with 4,000 IU of oral vitamin D3 daily.
4. The 25(OH)D3 increase achieved with the D3forME topical supplement patch will not differ between young and older adults.

To test these hypotheses, this research will be conducted in three stages:

Stage 1: Open Label Proof of Concept Pilot Study. This study will document safety and tolerability of daily D3forME topical supplement patches containing 4,000 IU of vitamin D3 in 15 healthy adult men and women.

The specific aims of this study are to:

1. Document the change in serum 25(OH)D3 with daily transdermal vitamin D3 dosing of 4,000 IU using the D3forME topical supplement patch.
2. Evaluate safety and skin tolerability of the D3forME topical supplement patch.

Stage 2: Efficacy study. In this randomized, double blind placebo controlled study of four months duration involving 40 healthy adult men and women (n = 20 per group) the specific aims are to:

1. Evaluate the safety and efficacy of daily D3forME topical supplement patches to increase serum 25(OH)D3.
2. Determine if the 25(OH)D3 increase achieved by 4,000 IU of daily D3forME topical supplement patches is superior to placebo.

Stage 3: Non-inferiority study. In this randomized, double blind placebo controlled study of six months duration involving 220 healthy adult men and women in two age cohorts, (18-40 years and 65-85 years), the specific aims are to:

1. Determine if the 25(OH)D3 increase achieved by 4,000 IU of daily D3forME topical supplement patches is not inferior to that achieved by 4,000 IU oral vitamin D3 supplementation.
2. Assess if the 25(OH)D3 increase achieved by daily D3forME topical supplement patches differs between young and old adults.

As an exploratory endpoint, the potential effect of body fat on response to daily D3forME topical supplement patches will be evaluated using DXA to measure body composition in the efficacy and non-inferiority studies (stages 2 and 3 above).

Open-label Proof of Concept Pilot Study. This open label study will evaluate the safety of a once daily D3forME topical supplement patches containing 4,000 IU of vitamin D3. Additionally, it will begin evaluating the efficacy of this approach on serum 25(OH)D3. This pilot study will include 15 healthy community dwelling men and women age 18-75 years without conditions contraindicating D supplementation or known skin conditions that could potentially interfere with cutaneous vitamin D3 delivery. Volunteers will be recruited from the Madison, WI area.

Stage 2: Randomized Double-blind, Placebo Controlled Efficacy Study: This study will include 40 adults (n = 20 in each group) using the same inclusion/exclusion criteria

Stage 3: Non-inferiority Study: This phase will include 220 adults randomly assigned to one of three treatment arms: n = 100 transdermal patch/placebo oral, n = 100 oral supplementation/placebo patch and n = 20 placebo oral and placebo patch) using the same inclusion/exclusion criteria as the noted above, except for age, which will be limited to 18-40 and 65-85. Additionally, each treatment arm will be equally divided into two cohorts, "young;" age 18-40 and "old;" age 65-85 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, community-dwelling ambulatory adults
* Able and willing to sign informed consent
* Age 18 to 75 years
* Baseline serum 25OHD concentration > 10 ng/mL and < 50 ng/mL
* Not pregnant
* Willing to not alter the amount of their baseline vitamin D supplementation during the course of this study
* Willing to utilize sunscreen of SPF-15 or higher when sun exposure for more than 15 minutes is expected

Exclusion Criteria:

* Current hypercalcemia (serum calcium > 10.5 mg/dl) or untreated primary hyperparathyroidism
* History of nephrolithiasis
* Baseline 24-hour urine calcium > 250 mg (female) or 300 mg (male)
* Known risk factors for hypercalcemia, e.g., malignancy, tuberculosis, sarcoidosis
* History of any form of cancer within the past five years with the exception of adequately treated squamous cell or basal cell skin carcinoma
* Renal failure; defined as a calculated creatinine clearance (using the Cockroft-Gault approach) of ≤ 35 ml/minute
* Severe end-organ disease, e.g., cardiovascular, hepatic, hematologic, pulmonary, etc., which might limit the ability to complete this study
* Treatment with any drug known to interfere with vitamin D metabolism, e.g., phenytoin, phenobarbital
* Known cutaneous sensitivity/allergy to tape or adhesives
* Known skin diseases, e.g., psoriasis, pemphigus, etc, which might alter transdermal vitamin D absorption
* Treatment with high dose vitamin D (≥ 50,000 IU weekly) or any active metabolites of vitamin D, e.g., calcitriol, within six months of screening
* Use of tanning beds or salons or unwillingness to utilize sunscreen during periods of sun exposure of 15 minutes or longer
* Planned trips/vacations likely to be associated with substantial amounts of sun exposure during the course of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Serum 25(OH)D | Change from baseline at 6 months
Serum 25 OHD | Change from baseline at 30 days
Serum 25(OH)D | Change from baseline at 4 months

SECONDARY OUTCOMES:
Skin Erythema | For Pilot up to 30 days, For Efficacy up to 4 months, and For non-inferiority up to 6 months
  Evaluate safety and skin tolerability of the D3forME topical supplement patch.

OTHER OUTCOMES:
Body Fat | During only the 2 and 3 phases, only at baseline visit.
  As an exploratory endpoint, the potential effect of body fat on response to daily D3forME topical supplement patches will be evaluated using DXA to measure body composition in the efficacy and non-inferiority studies.
Serum Calcium | For Pilot up to 30 days, For Efficacy up to 4 months, and For non-inferiority up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Osteoporosis Clinical Research Program, Madison, Wisconsin, United States